CLINICAL TRIAL: NCT01540032
Title: Low Salicylate Diet in Aspirin Exacerbated Respiratory Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AERD-01
Record Dates: First submitted 2012-02-09; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Aspirin Exacerbated Respiratory Disease; Samter's Triad

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
  Interventions: Behavioral: Normal diet
- Diet (Experimental)
  Interventions: Behavioral: Low salicylate diet

INTERVENTIONS:
Behavioral: Low salicylate diet — Patients will avoid foods from the 'high salicylate' group completely. They can eat foods from the 'low salicylate' group freely and just eat foods from the medium group occasionally, and not in large amounts.
  Arms: Diet
Behavioral: Normal diet — Patients will eat their usual diet.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether a low salicylate diet will improve the quality of life of patients with Aspirin Exacerbated Respiratory Disease (AERD).

DETAILED DESCRIPTION:
Aspirin-exacerbated respiratory disease (AERD) is clinically diagnosed in patients who suffer from allergy to aspirin, asthma, nasal polyps, and chronic sinusitis. Patients with AERD are often resistant to medical management of nasal polyps, and require multiple endoscopic sinus surgeries to manage recurrences of nasal polyps. Control of AERD can be obtained through aspirin desensitization, which consists of taking aspirin every day. However, there are substantial risks and adverse side effects to taking moderate amounts of aspirin daily. Furthermore, patients experience progressively worsening nasal and respiratory disease even with complete avoidance of aspirin and other NSAIDs.

The active and major component in aspirin/NSAIDs is salicylate, which is also found naturally in some foods. Diet modification is a cost-effective intervention that has the potential to provide long-term remission of AERD. Our study will evaluate whether a low salicylate diet, which is a more cost effective and benign intervention with minimal risks, will improve nasal, sinus or respiratory symptoms, such as congestion, sinusitis, smell, or asthma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AERD

Exclusion Criteria:

* Recent use of Prednisone or other systemic steroid (greater than three (3) doses in past three (3) months). This does not include the use of nasal steroids.
* Endoscopic sinus surgery / polypectomy within the past six (6) months
* Other significant systemic disease or immunocompromised state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Change in SNOT-22 scores from Baseline | 6 weeks and 12 weeks
  As this is a crossover study, all participants will complete the SNOT-22 questionnaire at the beginning of the study. After 6 weeks of their assigned diet (normal vs low salicylate), they will complete the SNOT-22 questionnaire to see if there are any differences in subjective nasal and sinus symptoms. After 6 weeks, the participants cross over to the other diet and they will complete the SNOT-22 questionnaire again in another 6 weeks when the study ends.

SECONDARY OUTCOMES:
Change in Lund-Kennedy Endoscopic Score from Baseline | 6 weeks and 12 weeks
  As this is a crossover study, all participants will be evaluated for the Lund-Kennedy Endoscopic Score at the beginning of the study. After 6 weeks of their assigned diet (normal vs low salicylate), they will be re-evaluated in clinic to see if there are any differences in endoscopy findings. After 6 weeks, the participants cross over to the other diet and they will have a final endoscopic evaluation in another 6 weeks when the study ends.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Health Care, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario